CLINICAL TRIAL: NCT01058356
Title: Effect of Probiotic Lactobacilli (Lacidofil Cap®) for the Prevention of Antibiotic-Associated Diarrhea: Prospective, Randomized Double-blind, Multicenter Study
Brief Title: Effect of Probiotic Lactobacilli (Lacidofil Cap®) for the Prevention of Antibiotic-Associated Diarrhea
Status: Completed | Type: Observational
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: NAM, Bong kil/ CEO & President, Pharmbio Korea
Other Study IDs: KASID_lacidofil_1
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Antibiotics Associated Colitis; Pulmonary Infection
Keywords: antibiotics associated colitis; lactobacilli; probiotics; prevention; pulmonary infection; Prevention of antibiotics associated colitis; the role of probiotics for prevention of antibiotics associated colitis; the lactobacilli effect for antibiotics associated colitis; antibiotic associated colitis on pulmonary infectious disease
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IBD research group in KASID: KASID is Korean Association Study of Intestinal Disease. It has several research group suh as inflammatory bowel disease (IBD) research group.

SUMMARY:
Antibiotic-Associated Diarrhea (AAD) is a common complication of antibiotic use. The frequency of AAD can be high (26 - 60%) or moderate (13-29%) during hospital outbreaks and is relatively infrequent in outpatients. The risk factors for AAD include broad-spectrum antibiotics, host factors (age, health status, and gender), hospitalization period and exposure to nosocomial pathogens. AAD occurs 2-8 weeks after exposure to antibiotics as a result of disrupting normal intestinal microflora. One of the roles of normal intestinal microflora is to act as a protective barrier that resists the colonization of intestinal pathogens. These patients are susceptible to infection by opportunistic pathogens without this protective barrier. Probiotic therapy is suited to AAD and Clostridium difficile disease. Probiotics assist in reestablishing the disrupted intestinal microflora, enhancing immune responses and clearing pathogens and their toxins from the host. Studies using probiotics have been reported for the past twenty-eight years (1977~2005), but the studies have been variable in trial designs and types of probiotics, had differing doses and durations of treatment, and thus have yielded controversial results. The investigators will conduct a multi-center, randomized, placebo-controlled, double-blind trial to assess the efficacy of the probiotic Lactobacilli (Lacidofil cap®) for the prevention of AAD in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18
* Patients with respiratory tract infection who are receiving an oral or injection antibiotics.
* Signed informed consent form prior to inclusion in the study.
* Patients who begin receiving antibiotics within 48 hours before enrollment in this study.

Exclusion Criteria:

* Diagnosed Clostridium difficile colitis within the last 3 months
* Patients with tube feeding, ileostomy or colostomy
* Patients with basal diarrheal disease; acute enteritis, chronic diarrhea such as inflammatory bowel disease (IBD) etc, radiation enteritis, ischemic colitis and diarrhea caused by carcinoids etc.
* Patients receiving other probiotics during the last 15 days
* Patients treated with immunosuppressant drugs or immune deficiency patients
* Patients with radiotherapy and chemotherapy treatment for cancer.
* Patients treated with antidiarrheal, antispasmodic or motility agents for other diseases.
* Pregnant/Lactating women
* Patients with gastrointestinal (GI) surgery during the last 3 months.
* A history of hypersensitivity to cephalosporins, penicillin or clavulanic acid.
* Patients with verified diabetic autonomic neuropathy.
* Patients with organ transplants.
* Patients with underlying conditions or diseases which, in the opinion of the investigator, are unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory tract infection who begin receiving antibiotic therapy (both hospitalized patients and out-patients)
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Ae Jung, MD, PhD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- KASID IBD Research Group, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2008 to November 2009, medical clinic
Pre-assignment Details: Patients who begin receiving antibiotics prior to 48 hours before enrollment in this study
Groups:
- Lacidofil Capsule Versus Placebo Drug: Lacidofil capsule: Lactobacillus rhamnosus R0011‧Lactobacillus acidophilus R0052 bacterial culture (2x109), maltodextrin, Mg stearate, ascorbic acid (1 capsule twice a day for 14 days) Placebo drug: maltodextrin, Mg stearate, ascorbic acid
  (1 capsule twice a day for 14 days)
Period: Overall Study
Arm/Group | Lacidofil Capsule Versus Placebo Drug
Started | 214
Completed | 172
Not Completed | 42
Not completed — Adverse Event | 5
Not completed — Administration of contraindicated drugs | 12
Not completed — Withdrawal by Subject | 21
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lacidofil Capsule Versus Placebo Drug
Number analyzed (Participants) | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 112
  >=65 years | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 60.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 132
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 214

OUTCOME MEASURES:

1. Primary Outcome: Presence of AAD
Description: AAD defined as: Watery stools more than 3 times per day for at least 2 days.
Time Frame: Up to 14 days
Measure: Number; unit: participants
Arm/Group | Lacidofil Capsule Versus Placebo Drug
Number analyzed (Participants) | 214
participants | 12
Statistical Analysis 1: Comparison: Lacidofil Capsule Versus Placebo Drug; Null hypothesis: The efficay of the probiotic Lactobacilli (Lacidofil cap®) for the prevention of AAD in adults is not different form the placebo group in multi-center, randomized, placebo-controlled, double-blind trial. Power calculation: The assumption of sample size calculation: difference 18% (8% : 26%) α: 0.05, statistical power: 90%, two sided difference: 18% Compliance: 80% - Unadjusted sample size (N=200) 180 + 10(%) drop out = 180 + 180/ (1-0.1)2 = 222.2 Total 220 subjects; Test type: Superiority or Other; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.17 to 4.15], Standard Error of Mean 0.40

2. Secondary Outcome: Presence of Bowel Habit Change (Watery Stools More Than 2 Times Per Day for at Least 2 Days)
Time Frame: Up to14 days
Measure: Number; unit: participants
Arm/Group | Lacidofil Capsule Versus Placebo Drug
Number analyzed (Participants) | 214
participants | 25
Statistical Analysis 1: Comparison: Lacidofil Capsule Versus Placebo Drug; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.18 to 1.55], Standard Error of Mean 0.27

ADVERSE EVENTS:
Arm/Group | Lacidofil Capsule Versus Placebo Drug
Serious Adverse Events (participants affected / at risk) | 0/214
Other Adverse Events (participants affected / at risk) | 0/214

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No